CLINICAL TRIAL: NCT00320320
Title: A Pilot Phase II Trial of Irinotecan Discontinuation and Reintroduction in Patients With Previously Untreated Advanced Colorectal Cancer
Brief Title: Irinotecan Discontinuation and Reintroduction for Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Gachon University Gil Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMO-GI-53
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal Neoplasms; Metastases
Keywords: No prior chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Irinotecan

SUMMARY:
The purpose of this study is to evaluate the feasibility and efficacy of first-line FOLFIRI discontinuation after initial 8 cycles and reintroduction after progression.

DETAILED DESCRIPTION:
For medically-fit patients with advanced colorectal cancer, the current standard approach is chemotherapy with FOLFIRI or FOLFOX. Although a strategy of using sequential 5-FU, irinotecan and oxaliplatin has been thought to maximize overall survival in such patients, significant toxicity remains a problem. It has been suggested feasible that chemotherapy can be discontinued after 2-3 months and restart same treatment on progression in patients with chemosensitive colorectal cancer. Thus we designed this pilot phase II study to evaluate the feasibility and efficacy of first-line FOLFIRI discontinuation after initial 8 cycles and reintroduction after progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of colon and rectum
* No prior chemotherapy or only adjuvant chemotherapy and/or radiotherapy
* Advanced, metastatic or recurrent not amenable to curative local therapy
* Measurable lesion(s)
* ECOG performance status 0 to 2
* Normal marrow, hepatic and renal function
* Provision of written informed consent

Exclusion Criteria:

* Active infection and/or severe comorbidity
* Known history of anaphylaxis of any origin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2005-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Response rate after FOLFIRI reintroduction

SECONDARY OUTCOMES:
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Gachon University Gil Medical Center, Incheon, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea